CLINICAL TRIAL: NCT04134416
Title: Effects of Combining Donepezil, Intensive Language Rehabilitation and Transcranial Direct Current Stimulation on Language Recovery and Brain Reorganization in Chronic Post-stroke Aphasia
Brief Title: Brain Correlates of Multimodal Rehabilitation in Chronic Post-stroke Aphasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Marcelo Luis Berthier, Full Professor, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIM-DON-2017-01
Record Dates: First submitted 2019-10-16; First posted 2019-10-22 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Aphasia; Stroke
Keywords: Aphasia; Stroke; Rehabilitation; Non-invasive brain stimulation; Cognitive enhancing drug; Intensive Language-Action Therapy
MeSH Terms: conditions — Aphasia; Stroke | interventions — Donepezil; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an open label except for the tCDS treatment which is double blind (AtDCS vs shamtDCS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal transcranial direct current stimulation (Experimental): Transcortical direct current stimulation (tDCS) will be applied using a STARSTIM neurostimulation device (Neuroelectrics, Barcelona). Each participant will receive 10 20-minute sessions while receiving REGIAplus (online). Group 1 will receive active stimulation (anodal stimulation, A-tDCS).The active electrode will be placed in the region of the lower right frontal rotation and the reference electrode in the extraencephalic zone (left clavicle). Combined rehabilitation sessions (REGIAplus/tDCS) will be conducted, as indicated above, in weeks 9 and 10 of the trial.
  Interventions: Drug: Donepezil; Behavioral: Intensive-Language Action Therapy; Device: Transcranial direct current stimulation
- Sham transcranial direct current stimulation (Sham Comparator): Group 2 will receive sham stimulation (S-tDCS). In the sham stimulation, the same helmet and electrode that is used in the active stimulation will be placed but, in this case, we will apply only a slight current at the beginning and end of the session with the objective of simulating the effects that are experienced with the active stimulation without producing significant cortical stimulation. The active electrode will be placed in the region of the lower right frontal rotation and the reference electrode in the extraencephalic zone (left clavicle). Combined rehabilitation sessions (REGIAplus/tDCS) will be conducted, as indicated above, in weeks 9 and 10 of the assay.
  Interventions: Drug: Donepezil; Behavioral: Intensive-Language Action Therapy; Device: Transcranial direct current stimulation

INTERVENTIONS:
Drug: Donepezil — Donepezil shall be administered at the times stipulated in the study design as follows: one 5 mg tablet at night for 4 weeks and then one 10 mg tablet at night until the end of the trial (week 10).
Behavioral: Intensive-Language Action Therapy — All patients participating in the study will receive in weeks 9 and 10 daily three and a half hours of ILATplus therapy. This therapy consists of 30 minutes of specific repetition training (tailored and reinforced by the therapist) before starting with classic ILAT for 3 hours/day during 10 consecutive days.
Device: Transcranial direct current stimulation — Transcortical direct current stimulation (tDCS) will be applied using a STARSTIM neurostimulation device (Neuroelectrics, Barcelona). Each participant will receive either anodal or sham 20-minute sessions while receiving ILATplus. In the sham stimulation, the same helmet and electrode that is used in the active stimulation will be placed but, in this case, we will apply only a slight current at the beginning and end of the session with the objective of simulating the effects that are experienced with the active stimulation without producing significant cortical stimulation. The active electrode will be placed in the region of the lower right frontal rotation and the reference electrode in the extraencephalic zone (left clavicle). Combined rehabilitation sessions (ILATplus/tDCS) will be conducted, as indicated above, in weeks 9 and 10 of the trial.

SUMMARY:
Post-stroke aphasia (PSA), the partial or total loss of the ability to produce and/or understand language associated with stroke, is a highly prevalent and disabling disorder that negatively impacts the personal, social and working life of patients and families. Modern theory-based language therapies (LT) with proved efficacy in chronic PSA are brief (weeks), intensive, and oriented to specific domains (e.g., anomia). However, in order to maximize therapeutic benefits, it becomes essential to implement complementary strategies that boost gains in language, communication and behaviour and also to identify predictors of treatment response (demographics, anatomical) that enable to customize interventions adjusting them to each profile (linguistic deficits, brain structure and connectivity). Our group has repeatedly shown that LT combined with cognitive enhancing drugs (CED) (e.g., Donepezil and Memantine) are safe and promote better outcomes that when these interventions are administered separately. Moreover, non-invasive brain stimulation techniques (NIBS), such as transcranial direct current stimulation (tDCS), are also emerging as a promising treatment option for chronic PSA. However, is still unknown whether or not treatments that combine several biological strategies aid to improve outcomes further. Brain changes induced by these interventions and the premorbid characteristic of a "good responder" are also unknown. The aims of this clinical trial are: (1) Study the efficacy of combined treatments in a sample of patients with chronic PSA (n = 40); (2) Document with multimodal neuroimaging the functional and connectivity changes (neuroplasticity) promoted by these interventions; and (3) Identify linguistic, cognitive and behavioural variables that may predict outcomes for each intervention.

DETAILED DESCRIPTION:
Aphasia is a devastating disorder involving total or partial loss of language. It can affect all communicative, expressive, and receptive modalities, including language production, comprehension, reading, writing, and the ability to gesture. Stroke is the most common cause of aphasia and its incidence is very high in Europe, varying between 318 and 372 cases in men and between 195 and 240 in women per 100,000 inhabitants. In Spain it is the second cause of death and the first in women, affecting approximately 130,000 people every year. Between 21 and 38% of these cases present post-stroke aphasia (PSA) in the acute stage. PSA is associated with high morbidity and mortality, and only 20% of those affected recover spontaneously. Consequently, PSA is very frequent and evolves to chronicity in most patients. There are different subtypes of aphasia depending on the linguistic profile. A distinction is made between aphasia with preserved repetition and aphasia with altered repetition. The first group includes transcortical aphasias (sensory, motor and mixed) and anomic aphasias, and the second, in order of severity, global aphasias, Wernicke aphasias, Broca aphasias, and Conduction Aphasias (CA). The latter group is associated with perisylvian lesions and are most frequent (>80% of cases). Aphasias in the first 2-3 months tend to evolve into less severe profiles, so that Broca and Wernicke aphasias can, in chronic stages, progress to CA.

Aphasia has a negative impact on the affected person and their family members, reducing work, personal, affective and social life. It is accompanied by high health and social expenditure, since one third of patients are under 65 years of age and cannot return to work due to the inability to communicate. For this reason, the implementation of strategies aimed at improving aphasia, communication, associated emotional disorders and the quality of life of patients and carers is crucial to achieve autonomy, allowing them to return to work and prevent additional cognitive and affective impairment. Currently, the most popular PSA rehabilitation therapies are: speech rehabilitation therapies, drugs and, more recently, non-invasive neurostimulation techniques.

1. Speech therapies Speech therapy is the treatment of choice in aphasia. The most commonly used is conventional or standard therapy where a specific strategy (description of pictures, repetition of words or phrases, answers to questions) is employed depending on the patient's deficits. They are usually applied 2 or 3 times a week with a duration of 30-45 minutes per session. However, some of the problems with these therapies are their prolonged duration (several years) and, consequently, their high cost, which limits their applicability in Public Health Services. In addition, the logistical limitations (difficulty of transport, shortage of staff) of the treatment centres prevent the administration of the minimum of 2 hours per week of therapy required to obtain clinically relevant benefits. On the other hand, the benefits obtained are insufficient and the progress made decreases once the treatment has been abandoned. For this reason, during the last two decades, speech therapies have been designed in which short (2 weeks) but very intensive (3 hours per day) rehabilitation exercises based on neuroscientific evidence are applied which effectively solve the limitations of traditional therapies. In this sense, Intensive Language-Action Therapy (ILAT) administered for two consecutive weeks (3 hours/day for 2 weeks - 30 hours of treatment -) has gained worldwide acceptance as it is significantly more effective than traditional rehabilitation techniques even when the total therapy time (2 hours/week for 15 weeks - 30 hours of treatment) is the same. In addition, the benefits achieved with ILAT in 2 weeks are maintained for 6 months after completion of treatment. ILAT is a group rehabilitation therapy (2 or 3 participants) that employs a play dynamic among participants, and its ILAT-plus modality also reinforces the training of specific language skills (e.g., repetition).
2. Pharmacological interventions LT is effective in the PSA, even in chronic stages (> 6 months after stroke). However, in many patients with moderate and severe aphasia the benefits of LT are limited (e.g., partial recovery of verbal fluency and auditory comprehension).These limitations have led to the use of other, more effective interventions to treat PSA. Several clinical trials in patients with acute and chronic PSAs conducted in the last decade have shown that the benefits achieved with rehabilitation can be significantly increased when these therapies are combined with drugs. Several pharmacological agents (Levodopa, Bromocriptine, Piracetam, Amantadine, Dexamfetamine, and others) have been used with variable results. However, several controlled clinical trials have found significant improvements in production deficits, understanding, and in the overall severity of aphasia in patients with PSAs treated with Piracetam, Donepezil, Galantamine, or Memantine. In PSA rehabilitation, biological and behavioral treatments strengthen the activity of perilesional regions and brain areas that previously did not perform language functions, but that after stroke are recruited vicariously increasing the ability of language recovery in the patient. In the last decade, it has been shown that the acetylcholinesterase inhibitor (an enzyme that degrades acetylcholine) Donepezil, and the NMDA receptor antagonist Memantine (antidementia drugs with a good safety/tolerability profile) are more effective than placebo in the treatment of PSA, especially when these are prescribed in association with rehabilitation techniques based on neuroscientific evidence.
3. Neurostimulation Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that induces changes in the excitability of brain tissue by increasing (anodal stimulation, A-tDCS) or decreasing (cathodal stimulation, C-tDCS) the activity of nerve cells by applying weak electrical currents. The theoretical justification for the use of tDCS as an adjuvant technique in PSA rehabilitation is based on the fact that it modulates (increases or decreases) the rate of neuronal discharge, presumably through changes in the resting potential of the membrane, and thus facilitates or hinders the functioning of connections between neuronal groups. tDCS has been shown to be effective in a variety of neurological and psychiatric disorders and has several advantages over other stimulation techniques, e.g. transcranial magnetic stimulation: better safety profile, easy to use, well tolerated by patients and better cost-benefit ratio. Increasingly, studies indicate that tDCS has beneficial effects on language deficits (verbal fluency, naming, grammatical decision) in people with PSA. In addition, when applied in conjunction with ST, it enhances the benefits obtained in PSA. Benefits have been described in patients with PSA using varied stimulation parameters (intensity, type, duration, brain area), each with different theoretical justification. The main modalities are (1) anodal stimulation (A-tDCS; excitatory) of perilesional areas with the aim of promoting the recovery of brain tissue surrounding the lesion; (2) cathodal stimulation (C-tDCS inhibitory stimulation of healthy regions interfering with recovery); (3) A-tDCS on areas of the healthy hemisphere to increase activity and facilitate the reorganization of functions that previously depended on injured areas of the left hemisphere. tDCS is a technique that has been shown to be effective, although more studies are needed leading to the identification of the most suitable stimulation parameters, the location-extent of the lesion, the previous brain structure of each patient, and to determine the added value that this technique provides in combination therapies.

Justification and project contributions Intensive ST, neurostimulation and pharmacological interventions have independently been shown to be effective in the rehabilitation of PSA. Previous work indicates that combination therapies (ILAT and drug therapy) are superior to other treatment options as they enhance synergistic mechanisms that promote improved learning, language and functional communication in affected individuals. However, more research is needed to explore the benefits of combination therapies (e.g. Donepezil, ILAT and tDCS) and to identify the mechanisms and structures that are modulated by each of these rehabilitation therapies and that mediate recovery, with the aim of establishing response predictors.

The aim of the current project is to evaluate the efficacy of ILATplus (ILAT + repetition/imitation training) (3 hours/day for 2 consecutive weeks, total = 30 hours) combined with Donepezil and tDCS in the treatment of cognitive deficits in patients with chronic post-stroke aphasias, with a special emphasis on Conduction Aphasia (CA).

Through the use of different neuroimaging techniques, the investigators seek to identify anatomical and functional changes that are related to the benefits observed after interventions, and analyze the role of the uninjured (right) hemisphere in recovery. The analysis of behavioral and neuroimaging data will allow us to identify possible predictors (demographic, structural, functional) of response.

The investigators hope that the results derived from this clinical trial will have a positive impact reflected in several aspects. This study may show for the first time the potential superiority of combined therapies (ILATplus/Donepezil/tDCS) over other treatment options. The analysis of the results, in combination with the findings of previous studies will allow to optimize the rehabilitation of the PSA with short intensive group therapies (ILAT) and consequently, more ecological and less expensive compared to the current rehabilitation strategies that use prolonged therapies generally with little efficacy. In addition, the results of this study will make it possible to identify patients who will benefit from this type of intervention based on anatomical and demographic predictors of response to treatment, and thereby improve their success.

Finally, this project will be carried out by a multi-disciplinary group with extensive scientific and technical experience in this line of research. The methodology to be used, as well as the potential results, are based on the progress achieved by basic neuroscientific research with translational impact on the neurorehabilitation of language alterations associated with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Right handedness (80 point in the Edinburgh Handedness Inventory)
* Spanish as native language
* Single left-hemisphere stroke
* Diagnosis of aphasia established by a score in the Aphasia Quotient of the Spanish version of the Western Aphasia Battery (WAB) < 93.8 points.

Exclusion Criteria:

* Dysarthria without aphasia
* Multiple or bilateral injuries
* Increased risk of a new stroke or unstable neurological condition (e.g. transient ischemic attacks)
* History of severe psychiatric illness (schizophrenia, major depression, bipolar disorder, anxiety disorders)
* Alcohol and substance use or abuse
* Coexistence of aphasia with dementia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Western Aphasia Battery (WAB) | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess major clinical aspects of language function: information content, fluency, auditory comprehension, repetition and naming.
  Changes from Baseline in Western Aphasia Battery scores at 8, 10 and 26 weeks. Minimum and maximum values: 0-100 points. Higher scores mean better outcome.
Communicative Activity Log (CAL) | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess communicative behavior in the everyday life of patients. Changes from Baseline in CAL scores at 8, 10 and 26 weeks. Minimum and maximum values: 0-90 points (0-40 points for quality of communication; 0-40 points for amount of communication). Higher values mean better outcome.
Stroke Aphasia Depression Questionnaire (SADQ-10) | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess depressive symptomatology in persons with post-stroke aphasia. Changes from Baseline in SADQ-10 scores at 8, 10 and 26 weeks. Minimum and maximum scores: 1-30 points. Lower values mean better outcome.
Stroke and Aphasia Quality of Life Scale 39 (SAQOL-39) | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess Quality of Life in persons with post-stroke aphasia. Changes from Baseline in SAQOL-39 scores at 8, 10 and 26 weeks. Minimum and maximum scores: 1-85 (Physical scale); 1-35 (Communication scale); 1-55 (Psychosocial scale); 1-20 (Vitality scale); 1-5 (Total mean scale).
  Higher values mean better outcome.

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE) | Each participant will be evaluated at week 0 (baseline).
  To assess cognitive impairment in persons with post-stroke aphasia. Minimum and maximum scores: 1-30 points. Higher values mean better outcome.
Trail-Making Test, parts A & B (TMT) | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess executive functions in individuals affected by post-stroke aphasia. Changes from Baseline in TMT scores at 8, 10 and 26 weeks. The participant has to finish both parts as quickly as possible, with the time taken to complete the test being used as the primary performance metric. Lower completion time means better outcome.
Digit Span Test from the Wechsler Adult Intelligence Scale (WAIS) | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess immediate memory in persons with post-stroke aphasia. Changes from Baseline in Digit scores at 8, 10 and 26 weeks. Minimum and maximum scores: 3-9. Higher values mean better outcome.
Attention Network Test (ANT). | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess three attentional networks: alerting, orienting, and executive control in in persons with post-stroke aphasia.
  Changes from Baseline in ANT scores at 8, 10 and 26 weeks. Efficiency of the alerting network is examined by changes in Reaction Time (RT) resulting from a warning signal. Efficiency of orienting is examined by changes in RT that accompany cues indicating where the target will occur. The efficiency of the executive network is examined by requiring the subject to respond by pressing two keys indicating the direction (left or right) of a central arrow surrounded by congruent, incongruent or neutral flankers.
  Lower reaction time and higher congruent responses mean better outcome.
Raven´s Colored Progressive Matrices (RPM), set A, B & AB | Each participant will be evaluated at week 0 (baseline).
  To assess abstract reasoning in persons with post-stroke aphasia. Evaluation at baseline. Minimum and maximum score: 0-36. Higher scores mean better outcome.
Cognitive Reserve Questionnaire. | Each participant will be evaluated at week 0 (baseline)
  To assess the cognitive reserve of persons with post-stroke aphasia. Evaluation at baseline. Minimum and maximum scores: 0-25. Higher values mean better outcome.
Hospital Anxiety and Depression Scale (HADS). | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess depressive and anxious symptomatology in persons with post-stroke aphasia.
  Changes from Baseline in HADS scores at 8, 10 and 26 weeks. Minimum and maximum scores: 0-21 points (Anxiety scale); 0-21 points (Depression scale). Lower values mean better outcome.
Visual Dynamic Analogue Scale (D-VAMS). | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess mood in persons with post-stroke aphasia. Changes from Baseline in D-VAMS scores at 8, 10 and 26 weeks. Minimum and maximum score: 0-100 points. Higher values mean better outcome.
Neuropsychiatric Inventory (NPI). | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess neuropsychiatric symptomatology in persons with post-stroke aphasia. Changes from Baseline in NPI scores at 8, 10 and 26 weeks. Minimum and maximum scores: 0-12 points for each subscale. Score obtained by multiplying frequency*severity scores. No total score available. Lower values mean better outcome.
Starkstein Apathy Scale (SAS). | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess apathy in persons with post-stroke aphasia. Changes from Baseline in SAS scores at 8, 10 and 26 weeks. Minimum and maximum scores: 0-42 points. Lower values mean better outcome.
Catastrophic Reaction Scale (CRS) | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess catastrophic reactions in persons with post-stroke aphasia. Changes from Baseline in CRS scores at 8, 10 and 26 weeks. Minimum and maximum scores: 0-33 points. Lower values mean better outcome.
Neurobehavioral Change after Aphasia Scale (experimental test). | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess personality changes in persons with post-stroke. Changes from Baseline scores at 8, 10 and 26 weeks. Minimum and maximum scores: 1-7 points for each subscale. Higher values mean better outcome.
Barthel Index (IB) | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess functional independence in persons with post-stroke aphasia. Changes from Baseline in functional independence scores at 8, 10 and 26 weeks. Minimum and maximum scores: 0-100 points. Higher values mean better outcome.
Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26.
  To rule out dementia in persons with post-stroke aphasia. Changes from Baseline in functional independence scores at 8, 10 and 26 weeks. Minimum and maximum scores: 26-130 points. Lower values mean better outcome.
Visual-analogue test assessing anosognosia for language impairment (VATA-L) | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26
  To screen for anosognosia for aphasia in persons with post-stroke aphasia. Changes from Baseline in anosognosia scores at 8,10 and 26 weeks. Minimum and maximum scores: 0-42. Lower values mean better outcome.
Communicative Effectiveness Index (CETI) | Each participant/ main carer will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess functional communication in persons with post-stroke aphasia. Changes from Baseline in functional communication scores at 8, 10 and 26 weeks. Minimum and maximum scores: 0-100. Higher values mean better outcome.
The Apraxia of Speech Rating Scale (ASRS). | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess and quantify the presence or absence, relative frequency, and severity of To rate apraxia of speech and its main characteristics in persons with post-stroke aphasia.
  Minimum and maximum scores: 0-4 points for each subscale. Lower values mean better outcome.
Corsi Block Tapping Test from the Wechsler Adult Intelligence Scale (WAIS) | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess visuo-spatial working memory in persons with post-stroke aphasia. Changes from Baseline in visual working memory scores at 8,10 and 26 weeks. Minimum and maximum scores: 3-9. Higher values mean better outcome.
Batería para la Evaluación de los Trastornos Afásicos (BETA). Battery for the Evaluation of Aphasia Disorders. Subscale 1,2,6,13,14,21 & 26. | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess linguistic abilities in persons with post-stroke aphasia. Subscales: 1,2,6,13,14,21 & 26 Changes from Baseline in linguistic abilities scores at 8,10 and 26 weeks. Minimum and maximum scores: 1-30. Higher values mean better outcome.
Queens List for the Repetition of Stimuli (experimental test) | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess linguistic abilities (repetition/naming) in individuals affected by post-stroke aphasia.
  Changes from Baseline in linguistic abilities scores at 8,10 and 26 weeks. Minimum and maximum scores: 1-48. Higher values mean better outcome.
Repetition of clichés and novel sentences (experimental test) | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess repetition of clichés and novel sentences in persons with post-stroke aphasia.
  Changes from Baseline in linguistic abilities scores at 8,10 and 26 weeks. Minimum and maximum scores: 0-40. Higher values mean better outcome.
Queens List for the Naming of Stimuli (experimental test) | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess linguistic abilities (repetition/naming) in individuals affected by post-stroke aphasia.
  Changes from Baseline in linguistic abilities scores at 8,10 and 26 weeks. Minimum and maximum scores: 1-48. Higher values mean better outcome.
Non-Verbal Oral Apraxia Screening Test (experimental test) | Each participant will be evaluated at week 0 (baseline), 8, 10 and 26.
  To assess non-verbal oral apraxia in individuals affected by post-stroke aphasia.
  Changes from Baseline (week 0) in oral apraxia scores at 8,10 and 26 weeks. Minimum and maximum scores: 0-32. Higher values mean better outcome.
Cognition test for Patients with Aphasia (experimental test) | Each participant will be evaluated at week 0 (baseline).
  To assess cognitive impairment in persons with post-stroke aphasia. Minimum and maximum scores: 1-30 points. Higher values mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo L Berthier, MD, PhD, Principal Investigator — University of Malaga, Spain
Locations (1):
- Centro de Investigaciones Medico-Sanitarias. University of Malaga, Málaga, Spain

REFERENCES:
- [Background] Berthier ML. Poststroke aphasia : epidemiology, pathophysiology and treatment. Drugs Aging. 2005;22(2):163-82. doi: 10.2165/00002512-200522020-00006. PMID 15733022
- [Background] Berthier ML, Garcia-Casares N, Walsh SF, Nabrozidis A, Ruiz de Mier RJ, Green C, Davila G, Gutierrez A, Pulvermuller F. Recovery from post-stroke aphasia: lessons from brain imaging and implications for rehabilitation and biological treatments. Discov Med. 2011 Oct;12(65):275-89. PMID 22031666
- [Background] Pulvermuller F, Berthier ML. Aphasia therapy on a neuroscience basis. Aphasiology. 2008 Jun;22(6):563-599. doi: 10.1080/02687030701612213. Epub 2008 May 21. PMID 18923644
- [Background] Berthier ML, Pulvermuller F. Neuroscience insights improve neurorehabilitation of poststroke aphasia. Nat Rev Neurol. 2011 Feb;7(2):86-97. doi: 10.1038/nrneurol.2010.201. PMID 21297651
- [Background] Berthier ML, Pulvermuller F, Davila G, Casares NG, Gutierrez A. Drug therapy of post-stroke aphasia: a review of current evidence. Neuropsychol Rev. 2011 Sep;21(3):302-17. doi: 10.1007/s11065-011-9177-7. Epub 2011 Aug 16. PMID 21845354
- [Background] Berthier ML, Green C, Higueras C, Fernandez I, Hinojosa J, Martin MC. A randomized, placebo-controlled study of donepezil in poststroke aphasia. Neurology. 2006 Nov 14;67(9):1687-9. doi: 10.1212/01.wnl.0000242626.69666.e2. PMID 17101908
- [Background] Berthier ML, Green C, Lara JP, Higueras C, Barbancho MA, Davila G, Pulvermuller F. Memantine and constraint-induced aphasia therapy in chronic poststroke aphasia. Ann Neurol. 2009 May;65(5):577-85. doi: 10.1002/ana.21597. PMID 19475666
- [Background] De-Torres I, Davila G, Berthier ML, Walsh SF, Moreno-Torres I, Ruiz-Cruces R. Repeating with the right hemisphere: reduced interactions between phonological and lexical-semantic systems in crossed aphasia? Front Hum Neurosci. 2013 Oct 18;7:675. doi: 10.3389/fnhum.2013.00675. eCollection 2013. PMID 24151460
- [Background] Torres-Prioris MJ, Lopez-Barroso D, Paredes-Pacheco J, Roe-Vellve N, Dawid-Milner MS, Berthier ML. Language as a Threat: Multimodal Evaluation and Interventions for Overwhelming Linguistic Anxiety in Severe Aphasia. Front Psychol. 2019 May 8;10:678. doi: 10.3389/fpsyg.2019.00678. eCollection 2019. PMID 31133908
- [Background] Mohr B, Stahl B, Berthier ML, Pulvermuller F. Intensive Communicative Therapy Reduces Symptoms of Depression in Chronic Nonfluent Aphasia. Neurorehabil Neural Repair. 2017 Dec;31(12):1053-1062. doi: 10.1177/1545968317744275. Epub 2017 Dec 1. PMID 29192534
- [Background] Berthier ML, De-Torres I, Paredes-Pacheco J, Roe-Vellve N, Thurnhofer-Hemsi K, Torres-Prioris MJ, Alfaro F, Moreno-Torres I, Lopez-Barroso D, Davila G. Cholinergic Potentiation and Audiovisual Repetition-Imitation Therapy Improve Speech Production and Communication Deficits in a Person with Crossed Aphasia by Inducing Structural Plasticity in White Matter Tracts. Front Hum Neurosci. 2017 Jun 14;11:304. doi: 10.3389/fnhum.2017.00304. eCollection 2017. PMID 28659776
- [Background] Barbancho MA, Berthier ML, Navas-Sanchez P, Davila G, Green-Heredia C, Garcia-Alberca JM, Ruiz-Cruces R, Lopez-Gonzalez MV, Dawid-Milner MS, Pulvermuller F, Lara JP. Bilateral brain reorganization with memantine and constraint-induced aphasia therapy in chronic post-stroke aphasia: An ERP study. Brain Lang. 2015 Jun-Jul;145-146:1-10. doi: 10.1016/j.bandl.2015.04.003. Epub 2015 Apr 29. PMID 25932618
- [Derived] Edelkraut L, Lopez-Barroso D, Torres-Prioris MJ, Starkstein SE, Jorge RE, Aloisi J, Berthier ML, Davila G. Spectrum of neuropsychiatric symptoms in chronic post-stroke aphasia. World J Psychiatry. 2022 Mar 19;12(3):450-469. doi: 10.5498/wjp.v12.i3.450. eCollection 2022 Mar 19. PMID 35433325
- See also: webiste of the university of Malaga, Spain — http://www.uma.es